CLINICAL TRIAL: NCT03004508
Title: Antioxidant Effect of Treatment With Ginkgo Biloba L. Leaf Extract (IDN 5933) on DNA Cell Maintenance and Genomic Stability: A Randomised Study Versus Placebo
Brief Title: Safety of Ginkgo Biloba Leaf Extract
Acronym: GiBiEx
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Indena S.p.A (Industry)
Responsible Party: Principal Investigator, Stefano Bonassi, Head, Clinical and Molecular Epidemiology, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDN5933
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Ginkgo Biloba Extract; Safety; Genomic Stability; DNA cell maintenance
MeSH Terms: conditions — Genomic Instability | interventions — Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gingko biloba Extract (Experimental)
  Interventions: Dietary Supplement: Gingko Biloba Extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Gingko Biloba Extract — 120mg/day, twice a day, 6 month
  Other Names: IDN 5933
  Arms: Gingko biloba Extract
Dietary Supplement: Placebo — 120mg/day, twice a day, 6 month
  Arms: Placebo

SUMMARY:
Primary objective: The primary objective of this study is to assess the effect of Ginkgo biloba L. leaf extract (IDN 5933) in comparison to placebo in human subjects treated at therapeutic doses for 6 months on the level of DNA damage and genomic instability, measured with the Comet Assay and the Micronucleus assay, respectively .

Secondary objective:

The secondary objective of this study is to provide a preliminary assessment of the safety of Ginkgo biloba L. leaf extract (IDN 5933) in human subjects treated at therapeutic doses in term of adverse drug reaction, hepatotoxicity, genotoxicity.

DETAILED DESCRIPTION:
The study will be a randomised clinical trial comparing subjects receiving twice-daily doses of either 120-mg of Ginkgo biloba L. leaf extract (IDN 5933) or placebo for a 6 months period.

Primary Endpoints:

* DNA Damage assessed with the Comet assay as proportion of DNA in the tail.
* Micronucleus frequency (MN) in peripheral blood lymphocytes (Frequency per 1000 binucleated cells).

Secondary Endpoints:

* Complete clinical assessment at the beginning and at the end of the study.
* Occurrence of Adverse drug reactions in individuals treated with GBE or placebo.
* Liver functions will be monitored according to biological laboratory examinations and clinical symptoms. A subgroup of individuals will be monitored also for genetic parameters concerning expression patterns of genes putatively associated to early events of HCC carcinogenesis Clinical and biological parameters will be measured in the study groups at the beginning (T0) and at the end of the study (T2).

ELIGIBILITY:
Inclusion Criteria:

* Male and female senior, residents of nursing homes, with no known clinically significant pathology as assessed by the investigator
* Life expectancy of greater than 1 year
* Subjects must have given written informed consent in accordance with ICH-GCP (International Conference on Harmonization - Good Clinical Practice) and local laws and regulations

To perform the experiment in a typical population treated with Ginkgo biloba L. leaf extract ( IDN 5933) the study will be performed among the residents of nursing homes among the structures of the San Raffaele network, i.e., The San Raffaele Montecompatri, the San Raffaele Rocca di Papa and the San Raffaele Sabaudia . The use of institutionalised subjects will allow a good compliance to the treatment, which will be administered by the nursing homes nurses.

Subjects meeting inclusion criteria and signing the informed consent will be randomised to receive 120-mg/twice per day of Ginkgo biloba L. leaf extract ( IDN 5933) or placebo.

Exclusion Criteria:

* Life expectancy of less than 1 year
* Treatment with anticoagulant and antiplatelet drugs in subjects with previous report of increased bleeding tendency
* Cognitive impairment
* Refuse to sign the informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
DNA Damage | through study completion, an average of 1 year
  DNA Damage assessed with the Comet assay as proportion of DNA in the tail
Micronucleus frequency | through study completion, an average of 1 year
  Micronucleus frequency (MN) in peripheral blood lymphocytes (Frequency per 1000 binucleated cells)

SECONDARY OUTCOMES:
Clinical assessment | through study completion, an average of 1 year
  Complete clinical assessment at the beginning and at the end of the study by physiological parameters
Liver functions | through study completion, an average of 1 year
  Liver functions will be monitored according to biological laboratory examinations and clinical symptoms
Gene Expression | A subgroup of individuals will be monitored also through study completion, an average of 1 year
  Expression patterns of genes putatively associated to early events of HCC carcinogenesis
Adverse drug reactions | through study completion, an average of 1 year
  Occurrence of Adverse drug reactions in individuals treated with GBE or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bonassi, PhD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele Pisana, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] National Toxicology Program. Toxicology and carcinogenesis studies of Ginkgo biloba extract (CAS No. 90045-36-6) in F344/N rats and B6C3F1/N mice (Gavage studies). Natl Toxicol Program Tech Rep Ser. 2013 Mar;(578):1-183. PMID 23652021
- [Result] Russo P, Frustaci A, Del Bufalo A, Fini M, Cesario A. Multitarget drugs of plants origin acting on Alzheimer's disease. Curr Med Chem. 2013;20(13):1686-93. doi: 10.2174/0929867311320130008. PMID 23410167
- [Result] Heinonen T, Gaus W. Cross matching observations on toxicological and clinical data for the assessment of tolerability and safety of Ginkgo biloba leaf extract. Toxicology. 2015 Jan 2;327:95-115. doi: 10.1016/j.tox.2014.10.013. Epub 2014 Nov 11. PMID 25446328
- [Result] Luo Y, Smith JV, Paramasivam V, Burdick A, Curry KJ, Buford JP, Khan I, Netzer WJ, Xu H, Butko P. Inhibition of amyloid-beta aggregation and caspase-3 activation by the Ginkgo biloba extract EGb761. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12197-202. doi: 10.1073/pnas.182425199. Epub 2002 Sep 4. PMID 12213959
- [Result] Bonassi S, Znaor A, Ceppi M, Lando C, Chang WP, Holland N, Kirsch-Volders M, Zeiger E, Ban S, Barale R, Bigatti MP, Bolognesi C, Cebulska-Wasilewska A, Fabianova E, Fucic A, Hagmar L, Joksic G, Martelli A, Migliore L, Mirkova E, Scarfi MR, Zijno A, Norppa H, Fenech M. An increased micronucleus frequency in peripheral blood lymphocytes predicts the risk of cancer in humans. Carcinogenesis. 2007 Mar;28(3):625-31. doi: 10.1093/carcin/bgl177. Epub 2006 Sep 14. PMID 16973674
- [Result] Collins A, Koppen G, Valdiglesias V, Dusinska M, Kruszewski M, Moller P, Rojas E, Dhawan A, Benzie I, Coskun E, Moretti M, Speit G, Bonassi S; ComNet project. The comet assay as a tool for human biomonitoring studies: the ComNet project. Mutat Res Rev Mutat Res. 2014 Jan-Mar;759:27-39. doi: 10.1016/j.mrrev.2013.10.001. Epub 2013 Oct 31. PMID 24184488
- [Derived] Bonassi S, Prinzi G, Lamonaca P, Russo P, Paximadas I, Rasoni G, Rossi R, Ruggi M, Malandrino S, Sanchez-Flores M, Valdiglesias V, Benassi B, Pacchierotti F, Villani P, Panatta M, Cordelli E. Clinical and genomic safety of treatment with Ginkgo biloba L. leaf extract (IDN 5933/Ginkgoselect(R)Plus) in elderly: a randomised placebo-controlled clinical trial [GiBiEx]. BMC Complement Altern Med. 2018 Jan 22;18(1):22. doi: 10.1186/s12906-018-2080-5. PMID 29357859